CLINICAL TRIAL: NCT05841706
Title: Open Label Randomized Trial of Blood Transfusions in Cancer Patients Following a Pancreatectomy: A Feasibility Study
Brief Title: Red Blood Cell Transfusion Thresholds for Improved Quality of Life for Patients Undergoing a Pancreatectomy for Pancreatic Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-001796
Record Dates: First submitted 2023-04-12; First posted 2023-05-03 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Resectable Pancreatic Carcinoma
Keywords: pancreatectomy, Transfusion
MeSH Terms: interventions — Hemoglobins; X-Rays; Specimen Handling; Pancreatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (Transfusion for Hgb less than 7 g/dL) (Experimental): Patients undergo red blood cell transfusion if Hgb is less than 7 g/dL while on study. Patients undergo CT scan, x ray imaging, and blood sample collection throughout the study.
  Interventions: Biological: Arm I Packed Red Blood Cell Transfusion (Hgb < 7 g/dL); Procedure: Computed Tomography; Procedure: X-Ray Imaging; Procedure: Biospecimen Collection; Other: Survey Administration; Procedure: Pancreatectomy
- Arm II (Transfusion for Hgb less than 9 g/dL) (Experimental): Patients undergo red blood cell transfusion if Hgb is less than 9 g/dL while on study. Patients undergo CT scan, x ray imaging, and blood sample collection throughout the study.
  Interventions: Biological: Arm II Packed Red Blood Cell Transfusion (Hgb < 9 g/dL); Procedure: Computed Tomography; Procedure: X-Ray Imaging; Procedure: Biospecimen Collection; Other: Survey Administration; Procedure: Pancreatectomy

INTERVENTIONS:
Biological: Arm I Packed Red Blood Cell Transfusion (Hgb < 7 g/dL) — Receive conservative transfusion strategy (Hgb < 7 g/dL)
  Other Names: PRBC Transfusion
  Arms: Arm I (Transfusion for Hgb less than 7 g/dL)
Biological: Arm II Packed Red Blood Cell Transfusion (Hgb < 9 g/dL) — Receive liberal transfusion strategy (Hgb < 9 g/dL)
  Other Names: PRBC Transfusion
  Arms: Arm II (Transfusion for Hgb less than 9 g/dL)
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT, CAT Scan, CAT scan, CAT Scan, Computed Axial Tomography, Computed Tomography, computed tomography
Procedure: X-Ray Imaging — Undergo x-ray imaging
  Other Names: Conventional X-Ray, Diagnostic Radiology, Medical Imaging, X-Ray, Radiographic Imaging, Radiography, RG, Static X-Ray, X-RAY, X-Ray, X-Ray, X-Ray, X-Ray
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection, Biological Sample Collection, Biospecimen Collected, Biospecimen Collection, Specimen Collection
Other: Survey Administration — Ancillary studies
Procedure: Pancreatectomy — surgical removal of all or part of pancreas

SUMMARY:
This clinical trial tests the the feasibility of testing a red blood cell transfusion threshold for improved quality of life for patients undergoing a pancreatectomy for pancreatic cancer. Pancreatectomy can be associated with significant blood loss. Blood loss can result in clinically important anemia causing fatigue. Pancreatic cancer itself can be associated with malnutrition and fatigue. Having a red blood cell transfusion threshold that results in a more liberal use of transfusions may improve quality of life for patients undergoing a pancreatectomy for pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. The primary objective for this pilot study is protocol adherence for the transfusion study we propose for pancreatectomy patients.

SECONDARY OBJECTIVES:

I. Determine the feasibility of collecting and processing of all data that will be collected in the full study.

II. Specific emphasis will be given to findings from Patient Reported Outcomes Measurement Information System (PROMIS)-29 to determine its sensitivity to changes in health related quality of life (HRQOL) that occur in the perioperative period after pancreatectomy.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo red blood cell transfusion if hemoglobin (Hgb) is less than 7 g/dL while on study.

ARM II: Patients undergo red blood cell transfusion if Hgb is less than 9 g/dL while on study.

Patients undergo computed tomography (CT) scan, x ray imaging, and blood sample collection throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >= 18 years of age at Visit 1
* Documentation of a pancreatic cancer diagnosis as evidenced by one or more clinical features meeting the following criteria:

  * CT evidence of a mass in the pancreas consistent with cancer
  * Tissue diagnosis of cancer either before surgery or from the resected specimen
  * Preoperative evaluation suggestive that pancreatic resection is feasible
* Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data
* Patients who are unable to receive or who refuse blood products
* Patients involved in an autologous pre-donation program
* Patients found to have metastatic disease upon entry into abdomen-having been randomized, these patients will be removed from the study and replaced with another patient
* Patients found to not have cancer during the operation- If the resected lesion proves not to be cancer, the patient will remain as an enrolled patient but not evaluable and replaced by another patient
* Established severe cardiovascular disease with estimated 5-year survival <10% based on Framingham risk score
* Unstable angina or recent myocardial infarction (MI)/stroke within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Rate of Protocol adherence | Up to 36 months post surgery
  Will be measured as the proportion of patients who are enrolled in the study and do not experience major protocol

SECONDARY OUTCOMES:
Health related quality of life | At preoperative visit, post operative period, months 1, 3, 6, 9, 12, 24, 27, 30, 33, 36
  Will be assessed by Patient Reported Outcomes Measurement Information System (PROMIS)-29 v2.1. PROMIS, uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. a higher T-score represents more of the concept being measured. For negatively-worded concepts like fatigue, a higher T-score represents greater fatigue and a lower T-score represents less fatigue. For positively-worded concepts like physical function, a higher T-score reflects higher (better) physical function and a lower T-score reflects lower (worse) physical function. For NIH Toolbox performance tests of cognitive, motor, and sensory function, a higher score indicates better performance.
Incidence of significant individual adverse events | Up to 36 months post operative
  Will include major adverse cardiovascular events (MACE), surgical site infection (SSI), surgical site occurrence (SSO), clinically-relevant postoperative pancreatic fistula (CR-POPF), hemorrhage, pneumonia, urinary tract infection (UTI), reoperation, readmission, and mortality. Safety and tolerability data will be summarized by treatment group. Adverse events will be tabulated by treatment group and will include the number of patients for whom the event occurred, the rate of occurrence, and the severity and relationship to study drug.
Length of stay in hospital and intensive care unit (ICU) | through study completion, an average of 1 year
Proportion of patients transfused | Up to hospital discharge or post operative day 28
Number of blood products received | Up to hospital discharge or post operative day 28

CONTACTS AND LOCATIONS:
Overall Officials: Edward Livingston, MD, Principal Investigator — University of California at Los Angeles
Locations (1):
- University of California at Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided